CLINICAL TRIAL: NCT02700256
Title: Electronic Patient-Reported Outcomes in Patients Recovering From Ambulatory Cancer Surgery: Measuring Early Postoperative Symptoms
Brief Title: Electronic Reporting of Symptoms After Surgery
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-315
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Patients Scheduled to Undergo Surgery on the Gynecology Service
Keywords: surgery; 15-315
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing a procedure: Patients will be asked to complete a baseline survey after enrollment. After surgery, enrollees who opt for the email/online access will receive an email upon discharge with a link to the WebCore site. Email will be sent at 9 am on postoperative day (POD) 2 to the email address the patient provided at consent. On post-operative days 2 through 6 the patient will be asked to complete a symptom inventory, they will receive an email with a link to the WebCore website, where they will be able to complete that day's survey. Enrollees who opt for the automated phone calls will complete their surveys via Interactive Voice Response (IVR), which will be automatically set-up to call the patient at 9 am on POD 2. Patients will complete phone surveys daily for 5 days. If the first phone call does not connect to the patient, a second phone call will be made at 10:00am. If the second call is unsuccessful a third & final call for that day will be placed at 11:00am.
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: survey — All patients will submit a baseline survey following enrollment onto study. After successful completion of the AXR or 24-hour discharge pathway, the consented patient will be contacted by email or telephone for 5 days following discharge from surgery.

SUMMARY:
The purpose of this pilot study is to find out if patients are willing to self-report symptoms in the first 5 days following discharge, or when they leave the hospital after "ambulatory surgery" ("ambulatory surgery" is when the patient has surgery and then goes home within 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* The patients must be undergoing surgery for an indication tracked within the Gynecologic AXR program or have an expected postoperative discharge within 24 hours of surgery. These surgical procedures typically include: minimally invasive hysterectomy or radical hysterectomy, salpingo-oophorectomies [mentioned above], and minimally invasive staging procedures.
* The patient must have a phone number or an email address.
* The patient must be willing to self-report postoperative symptoms over an automated phone system or via an online platform.
* The patient must speak and read fluent English.

Exclusion Criteria:

* Non-English speaking patients
* Patients unwilling to provide contact information (email or phone number)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo surgery on the Gynecology service through the AXR program or are discharged within 24-hours of surgery with internet access or a phone number will be recruited from the Rockefeller Outpatient Pavilion in the GYN Surgery Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
number of patients who respond to the survery | up to 5 days after surgery
  A patient will be deemed a "responder" if they complete at least 5 of the 8 symptom items on at least 3 days postoperatively. The symptom assessment method will be deemed successful if 32 of the 50 patients respond.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Zivanovic, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/